CLINICAL TRIAL: NCT03654235
Title: Pain Neuroscience Education and Physical Exercise Program in Patients With Chronic Back Pain. Intervention From Primary Care Physiotherapy Units
Brief Title: Pain Neuroscience Education and Physical Exercise Program in Chronic Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacion para la Investigacion y Formacion en Ciencias de la Salud (Other)
Collaborators: Castilla-León Health Service (Other); University of Valladolid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GRS 1396/A/16
Record Dates: First submitted 2018-08-24; First posted 2018-08-31 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Chronic Pain; Musculoskeletal Pain; Back Pain
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain; Back Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Patients Evaluator and Outcomes Assessor are masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNE and PE program (Experimental): Pain neuroscience education (Health education) and Physical exercise program.
  Interventions: Other: Health Education; Other: Physical exercise
- Usual care in Primary Care Physiotherapy (Active Comparator): Usual care in Primary Care Physiotherapy Units
  Interventions: Other: Usual care in Primary Care Physiotherapy Units

INTERVENTIONS:
Other: Health Education — 6 pain neuroscience education sessions (10 hours) and delivery of printed reinforcement material.
  Arms: PNE and PE program
Other: Physical exercise — Group physical exercise program (18 sessions; 3 sessions/week) leaded by a physiotherapist. It includes exercises to improve strength, coordination, balance and aerobic capacity. Work with double tasks, recreational activities to overcome kinesiophobia and activities to do at home are used in the program.
  Arms: PNE and PE program
Other: Usual care in Primary Care Physiotherapy Units — Treatment supported by the protocol of primary care of physiotherapy in the health service of Castilla y León that was in force at the time of the intervention.
  Patients receive 15 sessions of analgesic electrotherapy, thermotherapy and standardized physical exercise
  Arms: Usual care in Primary Care Physiotherapy

SUMMARY:
This study evaluates the effects of a pain neuroscience education (PNE) and physical exercise (PE) program in patients with chronic back pain. Half of participants receive PNE and PE program supervised by a physiotherapist and the other half receive usual physiotherapy care supported by physiotherapy protocols in primary care.

DETAILED DESCRIPTION:
Justification: Chronic musculoskeletal pain (CMP) affects more than 20% of the population, its prevalence is increasing, generating suffering and high health expenditure. The current knowledge of neurophysiology of pain shows that the painful experience in CMP is not necessarily associated with peripheral tissue damage and is due more to an alteration of central mechanisms of pain processing and to the dysfunction of endogenous pain inhibitory mechanisms. Physical exercise (PE) has been shown to be effective in CMP. Pain neuroscience education (PNE) improves the levels of pain catastrophism, Kinesiophobia, quality of life, disability and also modifies maladaptive cognitions that favour a painful response.

Objectives: To evaluate the efficacy of a PNE and PE in patients with chronic back pain (CBP). Changes in pain intensity, pain thresholds, Catastrophism, kinesiophobia, disability, central sensitization and quality of are measured.

Material and methods: Multicenter randomized clinical trial (RCT) with 170 patients. Intervention group receive 6 sessions of PNE and a 6 weeks PE program (18 sessions) aimed at improving functional capacity, neurogenesis and cerebral plasticity. Control group receive usual physiotherapy treatment (supported by the current protocols in Primary Care in the Health System of Castilla y León). The outcome variables are measured by Visual Analog Scale (EVA), Pressure Pain Threshold (PPT), Kinesiophobia Tampa Scale (TKS-11), Central Sensitization Questionnaire (CSC), Pain Catastrophism Questionnaire (CCD), disability (Roland-Morris), Quality of life (SF-36) and satisfaction (CSQ-8). An initial assessment, post-intervention (week 10), at six months and at year is performed. Patients Evaluator and Outcomes Assessor are masked.

Applicability of results: The proposed intervention is simple and reproducible. It can be performed in the Primary Care Physiotherapy Units. It requires few resources, and it can produce changes in pain intensity, functionality and quality of life of patients with CBP

ELIGIBILITY:
Inclusion Criteria:

* Nonspecific back pain of at least 6 months.
* Accept to participate in the study and sign the informed consent.

Exclusion Criteria:

* Oncological pain.
* Spine fracture or surgical intervention in last year.
* Neurological cognitive alteration that prevents understanding the contents of PNE program (In case of doubt, assesment with Minimental test)
* Motor control alteration that prevents the execution of the planned PE program (Minimum requirement: execution in normal time of the Timed Up and Go test)
* Pregnancy.
* Bladder or bowel incontinence.
* Saddle anesthesia.
* Patients presenting other clinical conditions that may aggravate chronic spinal pain (chronic fatigue syndrome, fibromyalgia and complex regional pain syndrome).
* Patients with associated pathologies that make it impossible to perform physical exercise program.
* Patients under treatment with alternative therapies.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Health-related Quality of Life at different time points | Change from baseline to post-treatment, to 6 months and at 12 months follow-up
  Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) V2. Spanish version. The SF-36 is a 36-item scale constructed to survey health status and quality of life. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary. Each scale is directly transformed into a 0-100 scale. Higher scores indicate better overall quality of life.

SECONDARY OUTCOMES:
Change in Pain assessment at different time points | Change from baseline to post-treatment, to 6 months and at 12 months follow-up
  Visual analog scale (VAS) scale. The VAS is a 100 mm long horizontal line ranging from '0: no pain at all' on one end to '100: worst pain imaginable' on the other end. Participants mark a point along the line that best represents the pain they are experiencing at that moment. A higher score indicates a higher level of pain.
Pressure pain threshold. | Change from baseline to post-treatment, to 6 months and at 12 months follow-up
  Pressure pain threshold (PPT). A digital pressure algometer is used at four standardized points to measure the pressure pain thresholds. Higher values represent a better tolerance to pressure pain.
Change in Pain Catastrophism at different time points | Change from baseline to post-treatment, to 6 months and at 12 months follow-up
  Pain catastrophizing scale (PCS). Spanish version. PCS is a short 13-item measure which evaluates the pain-related catastrophizing behaviours and cognitions of individuals. Score range from 0 - 52. A higher score indicates a higher level of catastrophism.
Change in Kinesiophobia at different time points | Change from baseline to post-treatment, to 6 months and at 12 months follow-up
  Tampa Scale of Kinesiophobia (TSK-11). Spanish version. TSK-11 is a self-report measure that contains 11 questions designed to assess a client's fear of movement and re-injury. Score range from 11 - 44. A higher score indicates a higher level of Kinesiophobia.
Change in Disability at different time points | Change from baseline to post-treatment, to 6 months and at 12 months follow-up
  Roland-Morris Disability Questionnaire (RMDQ). Spanish version. It is a self-administered disability questionnaire consisting of 24 questions that are specifically related to physical functions that may be affected by back pain. Score range from 0 - 24. A higher score indicates a higher level of Disability.
Change in Central sensitization levels at different time points | Change from baseline to post-treatment, to 6 months and at 12 months follow-up
  Central sensitization Inventory (CSI). Spanish version. Self-report instrument to detect the presence of central sensitization. It is a 25-item questionnaire that records the frequency of each symptom on a Likert scale from 0 (never) to 4 (always), resulting in a possible total score of 100. Higher scores are associated with higher levels of central sensitization.
Change in Drugs consumption | Change from baseline to post-treatment, to 6 months and at 12 months follow-up
  Record of consumption by types of drugs. Consumption is evaluated through a survey. The results are expressed in weekly doses per drug type.
Satisfaction survey. Satisfaction with the treatment | at 10 weeks
  Client Satisfaction Questionnaire (CSQ-8). Spanish version. It is is a self-report instrument used to assess satisfaction with health services and it is used to assess participant satisfaction with the treatment. Scores range from 8 - 32. Higher scores are associated with higher satisfaction.
Modifications of body mass index. | Change from baseline to post-treatment, to 6 months and at 12 months follow-up
  modification of the body mass index (BMI). Weight in Kg. and Height ill be combined to report BMI in kg/m^2.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A. Galán Martín, Principal Investigator — Castilla-León Health Service
Locations (1):
- Unidad de estrategias de Afrontamiento Activo para el dolor. Sacyl, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Galan-Martin MA, Montero-Cuadrado F, Lluch-Girbes E, Coca-Lopez MC, Mayo-Iscar A, Cuesta-Vargas A. Pain neuroscience education and physical exercise for patients with chronic spinal pain in primary healthcare: a randomised trial protocol. BMC Musculoskelet Disord. 2019 Nov 3;20(1):505. doi: 10.1186/s12891-019-2889-1. PMID 31679512